CLINICAL TRIAL: NCT05811793
Title: Efficacy and Safety of Superselective Cerebral Arterial Infusion of Bevacizumab Combined With Intrathecal Injection of Tislelizumab in the Treatment of Recurrent Glioblastoma
Brief Title: Efficacy and Safety of SCAI of Bevacizumab Combined With IC of Tislelizumab in the Treatment of Recurrent Glioblastoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-I-2023-016
Record Dates: First submitted 2023-03-21; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab arterial infusion combined with Tislelizumab intrathecal injection (Experimental): This is a prospective, interventional, multicenter Phase 2 trial for the treatment of patients with recurrent GBM who will receive Bevacizumab arterial infusion combined with Tislelizumab intrathecal injection. The study consists of two parts: the "arterial infusion part" in part 1, where each subject will receive 15 mg/Kg of Bevacizumab by cerebral arterial infusion over 15 minutes at a fixed time (d0, d30, d60); the infusion of 20% mannitol 12.5 ml over 120 seconds prior to the infusion of Bevacizumab; and the "intrathecal injection part" in part 2, where the subject will receive a fixed dose of intrathecal PD1 therapy (Tislelizumab 20 mg, d1, Q3W) intrathecal injection every 3 weeks for 6 cycles.
  Interventions: Drug: Tislelizumab and Bevacizumab

INTERVENTIONS:
Drug: Tislelizumab and Bevacizumab — Tislelizumab is a drug material authorized for marketing in China. Tislelizumab will be administered off-label in this study. Subjects with recurrent GBM will receive intrathecal tislelizumab every 3 weeks for six times. Intrathecal administration of Bevacizumab will be performed via Ommaya reservoir or intraventricular catheter.

SUMMARY:
To investigate the efficacy, safety and tolerability of superselective cerebral arterial infusion of Bevacizumab combined with intrathecal injection of Tislelizumab in the treatment of recurrent glioblastoma

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is a highly malignant intracranial tumor with a median survival of only about 15-17 months after standard treatment. Patients with GBM often experience disease recurrence, and once recurrence occurs, treatment options are very limited, with a median overall survival of only about 6 months. Results of a phase II clinical trial of nivolumab combined with standard or reduced-dose bevacizumab iv therapy for recurrent GBM showed that the median PFS for the two groups was 5.6 months vs. 4.6 months, respectively. The aim of this study is to improve the outcome of recurrent GBM patients by changing the route of administration of the two drugs, such as delivering Bevacizumab via intra-arterial infusion and administering PD-1 monoclonal antibodies via intrathecal injection.

ELIGIBILITY:
Inclusion Criteria:

* 1, 18 ≤ age ≤ 75 years. 2. Recurrent glioblastoma who failed first-line therapy, with no more than 3 prior episodes of disease progression and at least one confirmed and evaluable lesion.

  3. ECOG score 0-2 points, expected survival time ≥ 3 months; 4. Stable neurological symptoms for more than 7 days; 5. If the previous surgical resection interval is at least 4 weeks, after receiving chemotherapy for 3 weeks, after receiving radiotherapy including whole brain radiotherapy, stereotactic radiotherapy and other radiotherapy for 3 months, if receiving other intrathecal treatment drugs washout period of 7 days.

  6. Neutrophil count ≥ 1.5 × 10 ^ 9/L, hemoglobin ≥ 80 g/L, platelets ≥ 75 × 10 ^ 9/L.

  7. Prothrombin time/international normalized ratio and partial thromboplastin time ≤ 1.5 × upper limit of normal; 8. Total bilirubin ≤ 1.5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ×ULN, albumin ≥ 30 g/L, creatinine ≤ 2 × ULN, calculated creatinine clearance ≥ 50 mL/min, 24-hour urine creatinine clearance ≥ 50 mL/min; 9. subjects should agree to use adequate contraception from the first dose until 3 months after the last dose.

Exclusion Criteria:

* 1. Pregnant or lactating women. 2. Active infection requiring intravenous antibiotics requiring therapeutic anticoagulation with warfarin.

  3. History of allergy to monoclonal antibodies; 4. Use of non-tumor vaccines containing live viruses to prevent infectious diseases within 12 weeks before the study drug; 5. Subjects with serious medical, neurological or psychiatric disorders and judged to be unable to fully comply with study treatment or assessments; 6. Active infectious diseases within 7 days before starting the study drug; 7. Severe liver dysfunction (persistent grade 3 or greater liver adverse events) or known active chronic hepatitis, human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) test positive; 8. Patients with active autoimmune diseases requiring systemic treatment (i.e., the use of corticosteroids or immunosuppressive agents), except replacement therapy (e.g., thyroxine, insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency), allowing inhalation or local steroids and adrenal replacement dose > 10 mg daily prednisone equivalent, requiring long-term systemic corticosteroid therapy (> 10 mg prednisone or equivalent per day) or any other immunosuppressive therapy (including anti-TNF-a therapy); 9. Investigate the allergic history of drug ingredients; 10. Inadequate control of hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg (using antihypertensive drugs); 11. Any past history of hypertensive crisis or hypertensive encephalopathy; 12. New York Heart Association (NYHA) Class II or greater congestive heart failure; 13. History of myocardial infarction or unstable angina within 6 months prior to enrollment; 14. History of stroke or transient ischemic attack within 6 months prior to enrollment; 15. Severe vascular diseases (such as aortic aneurysm, aortic dissection); 16. Symptomatic peripheral vascular disease. 17. Evidence of bleeding diathesis or coagulopathy. 18. Major surgery, open biopsy or severe traumatic injury within 28 days prior to study enrollment, or major surgery is expected to be required during the course of the study.

  19. Core biopsy or other minor surgical procedures, excluding placement of vascular access devices, within 7 days prior to study enrollment.

  20. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to study entry; 21. Severe, non-healing wounds, ulcers or fractures. 22. Urine protein to creatinine ratio ≥ 1.0 or urine protein ≥ 2 +. 23. Subjects with high intracranial pressure who are not suitable for lumbar puncture, and the researchers believe that they are not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 10 approximately months
  PFS was defined as the time from random assignment until objective tumor progression (independent image committee assessment) or death (any cause)

SECONDARY OUTCOMES:
Objective Response Rate | Up to 10 approximately months
  ORR is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set.
Overall Survival | Up to 10 approximately months
  OS was defined as the time from random assignment until death (any cause) or censored at the last date of known survival.
Duration of Response | Up to 10 approximately months
  Time from the patient 's first assessment of clinical response to the first assessment of disease progression or death from any cause.
Safety and Tolerability | Up to 10 approximately months
  The safety endpoints will be assessed by a review of adverse events and serious adverse events according to CTCAE up to 10 approximately months after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Xingen Zhu, Dr., Principal Investigator — Second Affiliated Hospital of Nanchang University

IPD SHARING:
Plan to Share IPD: No